CLINICAL TRIAL: NCT04727762
Title: Population Impact on the Continued Use of the Mask Due to the Avoidance of COVID-19
Brief Title: Use of the Mask and Current Pandemic
Acronym: Mask
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Principal Investigator, University of Valencia
Other Study IDs: ID0031
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Face Mask Squeeze
Keywords: protection; SARS-CoV-2; cephalalgia; mastication; well-being
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Due to the continued use of the mask in order to prevent the spread of COVID-19, an impact on people is observed in different areas. The objective of our study was to collect impact aspects related to the continued use of the mask that may affect the quality of life of the population. For this, an observational study has been carried out that includes an interview with aspects related to headaches, problems in the temporomandibular joint, headache impact and quality of life.

DETAILED DESCRIPTION:
Introduction

Due to the continued use of the mask in order to prevent the spread of COVID-19, an impact on people is observed in different areas. The objective of our study was to collect impact aspects related to the continued use of the mask that may affect the quality of life of the population.

Material and methods

Diseny. For this, an observational study has been carried out that includes an interview with aspects related to headaches, problems in the temporomandibular joint, headache impact and quality of life.

Participants. Subjects of all ages from 18 years old will be recruited who use a mask daily for the avoidance of COVID-19 and with the ability to answer the questions and complete the questionnaires. The study will be carried out at the Faculty of Physiotherapy of the University of Valencia. The participants will sign an informed consent guaranteeing the confidentiality of the data. The study is approved by the ethics committee of our institution.

Outcomes. The sociodemographic characteristics and the use of the mask will be collected. Subsequently, the evaluation instruments without the use of a mask and with the use of the same in: Headache and the impact on headaches, pain related to temporomandibular joint and quality of life.

All data will be coded in a database and analyzed later.

ELIGIBILITY:
Inclusion Criteria:

* from 18 years old will be recruited who use a mask daily for the avoidance of COVID-19.
* that they use the face mask at least 2 hours a day
* with the ability to answer the questions and complete the questionnaires.

Exclusion Criteria:

* I do not use the mask
* institutionalized subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects of all ages from 18 years old will be recruited who use a mask daily for the avoidance of COVID-19 and with the ability to answer the questions and complete the questionnaires.
Sampling Method: Probability Sample
Enrollment: 542 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Headache | 1 day
  An ad hoc questionnaire will be carried out that includes a question about the existence of headache before and after the use of the mask with a dichotomous response (Yes, No) and another about the frequency of headache with the options of daily, weekly or monthly.
Pain Temporomandibular Joint | 1 day
  The ad hoc questionnaire will include two questions about the existence of joint discomfort in the TMJ before and after the use of the mask with a dichotomous response (Yes, No) and pain when chewing evaluated using the Visual Analog Scale (VAS).

SECONDARY OUTCOMES:
Headache Impact | 1 day
  Headache Impact Test-6 (HIT-6).To measure the impact of headache. The score is calculated as follows: never (6 points), few times (8 points), sometimes (10 points), very often (11 points) and always (13 points). With a total of 49 or less points is considered "little or no impact", between 50-55 "some impact", between 56-59 "significant impact" and 60 or more "very severe impact".
Influence on quality of life | 1 day
  Will be measured by Cantril Ladder of Life Scale (LADER). The Cantril Staircase (Cantril 1965), measures satisfaction with life. The subject is asked to imagine his life in the best possible way and to describe his hopes and wishes. You are then asked to imagine your future in the worst possible light, your fears and concerns associated with this outcome. Subsequently, the respondent is presented with an image consisting of a ladder numbered from zero to ten, where the top of the ladder represents the best possible life for the subject = 10 and the bottom of the ladder represents the worst possible life = 0.

CONTACTS AND LOCATIONS:
Overall Officials: Gemma V Espí-López, Principal Investigator — fisiotherapy
Locations (1):
- Gemma Victoria Espí-López, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No